CLINICAL TRIAL: NCT01374321
Title: Phase II, Multicenter, Randomized, Double-blind, Placebo Controlled Study to Assess Safety and Efficacy of TRO40303 for Reduction of Reperfusion Injury in Patients Undergoing Percutaneous Coronary Intervention for Acute Myocardial Infarction
Brief Title: Safety and Efficacy Study of TRO40303 for Reduction of Reperfusion Injury in Patients Undergoing Percutaneous Coronary Intervention for Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRO40303CLEQ1491-1
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Acute Myocardial Infarctus
MeSH Terms: interventions — 3,5-seco-4-norcholestan-5-one oxime-3-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TRO40303 (Experimental)
  Interventions: Drug: TRO40303

INTERVENTIONS:
Drug: TRO40303 — 6 mg/kg, peripheral IV, single dose just before balloon inflation, slow bolus (35ml/min)
  Arms: TRO40303
Drug: Placebo — single dose just before balloon inflation by slow bolus (35ml/min, peripheral IV)
  Arms: Placebo

SUMMARY:
Objectives of the phase 2 prospective, multicenter, randomized, double-blind, placebo-controlled study is to assess safety and efficacy of TRO40303 administered just before balloon inflation during percutaneous coronary intervention (PCI) for limitation of infarct size in patients treated for acute myocardial infarction (AMI).

The study is being conducted in 9 centres in Sweden, Denmark, Norway and France. One hundred eighty patients will be included. It will last one month per patient and its overall duration will be 11 months.

The efficacy will be assessed by infarct size expressed as area under the curve for creatine kinase and troponin I (blood sampling at D1, D2 and D3), and also evaluated by Cardiac Magnetic Resonance.

Safety will be assessed by

* clinic evaluation,
* blood samples (hematology, biochemistry, renal and hepatic function),
* Recording and follow-up of major adverse events occurring during the first 48h after reperfusion (death, heart failure, AMI, stroke, recurrent ischemia, the need for repeat revascularization, renal or hepatic, vascular complication and bleeding).
* ECG
* Recording cardiac events during one month after AMI
* Follow-up of global left ventricular function by Echocardiography at D3 and D30.

Demographic and medical history at inclusion and non-cardiac events occurring during the first 30 days will be recorded. TRO40303 plasma concentration will be assessed at 15 min, 6h, and 12h post the end of administration.

Sample size calculation assuming a reduction of 35% of the AUC for Troponin I release, for a statistical power of 85% and a probability of type I error of 0.05.

Main analysis: between-group comparisons of AUCs for serum troponin I and CK release will be performed using O'Brien's method for multiple endpoints testing.

Secondary analysis: comparisons of the CMR criteria described above will be performed using mixed model of ANCOVA.

All analyses will be performed on the Full Analysis Set and Per protocol populations.

Safety analysis: A comparison of the incidence of cumulative adverse clinical events between the groups will be performed by Fisher's exact tests.

Subjects will undergo primary PCI and receive concomitant medications according to current standard of care.

After coronary angiography is performed but just before balloon inflation is performed, patients who meet the enrollment criteria will be randomly assigned to either the control group or the TRO40303 group. Randomization is ensured by taking the treatment units in ascending and consecutive order in each strata (anterior/posterior as determined on ECG). Just before balloon inflation, ideally less than 5 minutes, and with a maximum of 15 minutes before balloon inflation and stenting, the patients in the TRO40303 group will receive an intravenous slow-bolus (35 mL/min) injection of 6 mg/kg of TRO40303 injected in peripheral IV. The patients in the control group will receive an equivalent volume of the placebo. Patients will be hospitalized for as long as there is a medical indication. CMR and echocardiography will accordingly be conducted as in/out patient between day 3 (ideally) and 5. A follow-up visit will be conducted one month after PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female with non childbearing potential patients
2. Age > 18 years old
3. First acute myocardial infarction
4. Occlusion should affect the following coronary arteries: LAD,or the dominant or balanced RCA, or the dominant or balanced LCx
5. Acute myocardial infarction defined as

   * nitrate resistant chest pain ≥ 30 min
   * ST elevation: New ST elevation at the J-point in two contiguous leads with the cut-off points: ≥ 2 mV in men or ≥ 0.15 mV in women in leads V2-V3 and/or ≥ O.1 mV in other leads
6. Presenting within 6h of onset of chest pain
7. Clinical decision to treat with percutaneous coronary intervention
8. Occlusion of culprit artery with a Thrombolysis In Myocardial Infarction (TIMI) flow grade 0-1 at time of admission and before percutaneous coronary intervention
9. Have signed an Informed Consent to participate to the trial before any study related procedure has been taken

Exclusion Criteria:

1. Cardiac arrest, ventricular fibrillation, cardiogenic shock, stent thrombosis, previous AMI, angina within 48h before admission, previous CABG, treatment with intravenous fibrinolytic therapy within the 72 hours to PCI
2. Atrial fibrillation (could confound CMR analysis)
3. Pace-maker
4. Concurrent inflammatory, infectious or malignant disease
5. Biliary obstruction or hepatic insufficiency at the time of inclusion in the study
6. Be possibly dependent on the Investigator or the Sponsor (eg including but not limited to affiliated employee)
7. Participated in any other investigational drug or therapy study with a non-approved medication, within the previous 3 months
8. Patient under guardianship
9. History of egg allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Infarct size expressed as area under the curve for Creatine kinase and Troponin I | Blood samples will be collected at admission and every 6 hours until 72h

SECONDARY OUTCOMES:
Infarct size evaluated by Cardiac Magnetic Resonance | A cardiac magnetic resonance between day 3 and Day 5 after balloon inflation

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, Pr, Principal Investigator — Ullevaal University Hospital
Locations (11):
- Denmark (2):
  - Aarhus University Hospital, Aalborg
  - Odense University Hospital, Odense
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital La Timone, Marseille
  - Hôpital Nord Marseille, Marseille
  - Hôpital Européen Georges Pompidou, Paris
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Larsen, Stavanger
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm

REFERENCES:
- [Derived] Nordlund D, Heiberg E, Carlsson M, Frund ET, Hoffmann P, Koul S, Atar D, Aletras AH, Erlinge D, Engblom H, Arheden H. Extent of Myocardium at Risk for Left Anterior Descending Artery, Right Coronary Artery, and Left Circumflex Artery Occlusion Depicted by Contrast-Enhanced Steady State Free Precession and T2-Weighted Short Tau Inversion Recovery Magnetic Resonance Imaging. Circ Cardiovasc Imaging. 2016 Jul;9(7):e004376. doi: 10.1161/CIRCIMAGING.115.004376. PMID 27412659
- [Derived] Engblom H, Tufvesson J, Jablonowski R, Carlsson M, Aletras AH, Hoffmann P, Jacquier A, Kober F, Metzler B, Erlinge D, Atar D, Arheden H, Heiberg E. A new automatic algorithm for quantification of myocardial infarction imaged by late gadolinium enhancement cardiovascular magnetic resonance: experimental validation and comparison to expert delineations in multi-center, multi-vendor patient data. J Cardiovasc Magn Reson. 2016 May 4;18(1):27. doi: 10.1186/s12968-016-0242-5. PMID 27145749
- [Derived] Tufvesson J, Carlsson M, Aletras AH, Engblom H, Deux JF, Koul S, Sorensson P, Pernow J, Atar D, Erlinge D, Arheden H, Heiberg E. Automatic segmentation of myocardium at risk from contrast enhanced SSFP CMR: validation against expert readers and SPECT. BMC Med Imaging. 2016 Mar 5;16:19. doi: 10.1186/s12880-016-0124-1. PMID 26946139